CLINICAL TRIAL: NCT03802123
Title: A Phase II, Open Label, Multi-Dose Study of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) for Positron Emission Tomography (PET/CT) in Patients With Selected Advanced or Metastatic Solid Malignancies Who Are Scheduled to Receive Standard-of-Care Immunotherapy Only, As Single Agent or in Combination
Brief Title: ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) for PET/CT in Patients With Metastatic Solid Tumors
Acronym: iCorrelate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: ImaginAb, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IAB-CD8-201
Record Dates: First submitted 2018-12-19; First posted 2019-01-14 (Actual); Results first posted 2024-07-09 (Actual); Last update posted 2024-07-09 (Actual); Status verified 2024-06

CONDITIONS: Positron-Emission Tomography; Metastatic Solid Tumors
Keywords: PET/CT; ⁸⁹Zr-Df-IAB22M2C; CD8; Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ⁸⁹Zr-Df-IAB22M2C Infusion (Experimental): A dose of 3 mCi (±20%) of ⁸⁹Zr-Df-IAB22M2C between 0.5 mg to 1.5 mg of API will be administered intravenously over 5-10 minutes, within one week prior to the onset of immunotherapy, and 5 to 6 weeks after start of IOT.
  Interventions: Drug: ⁸⁹Zr-Df-IAB22M2C

INTERVENTIONS:
Drug: ⁸⁹Zr-Df-IAB22M2C — ⁸⁹Zr-Df-IAB22M2C CD8 T cell tracer for Positron Emission Tomography (PET)

SUMMARY:
The purpose of this study is to evaluate the safety of repeat doses ⁸⁹Zr-Df-IAB22M2C and to establish the relationship between ⁸⁹Zr-Df-IAB22M2C PET/CT lesion uptake with CD8+ cells by immunohistochemical staining in patients with selected advanced and metastatic solid malignancies who are scheduled to receive standard of care immunotherapy. The study will also evaluate uptake of ⁸⁹Zr-Df-IAB22M2C by PET/CT in patients at baseline and on immunotherapy.

DETAILED DESCRIPTION:
After being informed about the study and potential risks, all patients giving written informed consent will be evaluated to determine eligibility for study entry. Up to 1 week prior to initiation of immunotherapy, patients will receive an injection of ⁸⁹Zr-Df-IAB22M2C (1.0 mCi) and will undergo PET/CT scanning to determine baseline uptake of ⁸⁹Zr-Df-IAB22M2C in tumor lesions and reference tissues. Patients will receive an additional injection of ⁸⁹Zr-Df-IAB22M2C (1.0 mCi) and PET/CT scan 4-6 weeks after starting immunotherapy (on-therapy) to evaluate uptake of ⁸⁹Zr-Df-IAB22M2C in tumor lesions and reference tissues, and to assess potential changes in uptake of ⁸⁹Zr-Df-IAB22M2C compared to the baseline scan.

ELIGIBILITY:
Inclusion Criteria:

Participants will be eligible for enrollment in the study only if they meet ALL of the following criteria:

1. 1. Patients with advanced or metastatic Melanoma, Non-Small Cell Lung Cancer, Renal Cell Carcinoma or Squamous Cell Carcinoma of the Head and Neck with at least one non-radiated lesion, who are scheduled to begin standard of care immunotherapy.
2. • At least 1 non radiated measurable lesion documented on CT/, MRI (per RECIST criteria 1.1) or are FDG avid on FDG-PET within 45 days prior to first 89Zr-Df-IAB22M2C (CD8 PET Tracer) infusion.
3. At least 1 non-cutaneous lesion that is accessible, per investigator's assessment, and eligible for biopsy. If only a single RECIST measurable lesion is present, investigator to determine if the tumor biopsy could interfere with RECIST assessments of response.
4. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2.
5. Meeting all clinical safety lab values per institution's standard of care, or Investigator's discretion, for patients receiving cancer treatment.
6. Age ≥ 18 years.
7. Ability to understand the purposes and risks of the trial and has signed an IRB-approved informed consent form.
8. Willingness and ability to comply with all protocol required procedures.
9. For men and women of child-producing potential, use of effective double barrier contraceptive methods during the study, up to 30 days after the last administration of the investigational product.

Exclusion Criteria:

Subjects will NOT be eligible for enrollment in the study if they meet ANY of the following criteria:

1. Serious nonmalignant disease or conditions that in the opinion of the investigator and/or ImaginAb could compromise protocol objectives.
2. Patients with a single RECIST measurable lesion, biopsy of which, per investigator's assessment, is likely to interfere with RECIST assessments of response.
3. Patients who have any splenic disorders, or had splenectomy, that in the opinion of the investigator and/or ImaginAb could compromise protocol objectives.
4. Pregnant women or nursing mothers.
5. 5. Life expectancy < 6 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2018-12-18 (Actual); Primary Completion 2021-10-19 (Actual); Study Completion 2022-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ron Korn, MD, PhD, Study Director — ImaginAb, Inc.
Locations (15):
- United States (15):
  - University of Alabama-Birmingham Hospital, Birmingham, Alabama
  - CARTI Cancer Center, Little Rock, Arkansas
  - City of Hope (City of Hope National Medical Center, City of Hope Medical Center), Duarte, California
  - Keck Hospital of USC, Los Angeles, California
  - LAC + USC Medical Center, Los Angeles, California
  - USC/Norris Comprehensive Cancer Center, Los Angeles, California
  - Hoag Memorial Hospital Presbyterian, Newport Beach, California
  - John Wayne Cancer Institute at Providence Saint John's Health Center, Santa Monica, California
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Dana-Farber Cancer Institute (DFCI), Boston, Massachusetts
  - Karmanos Cancer Institute, Detroit, Michigan
  - Washington University School of Medicine, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Pennsylvania, Perelman School of Medicine, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance/ University of Washington, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ⁸⁹Zr-Df-IAB22M2C Infusion: A dose of 3 mCi (±20%) or 1 mCi (±20%) of ⁸⁹Zr-Df-IAB22M2C at 1.5 mg of API will be administered intravenously over 5-10 minutes, within one week prior to the onset of immunotherapy, and 5 to 6 weeks after start of IOT.
  ⁸⁹Zr-Df-IAB22M2C: ⁸⁹Zr-Df-IAB22M2C CD8 T cell tracer for Positron Emission Tomography (PET)
Period: Overall Study
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Started | 52
Completed | 43
Not Completed | 9
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Subject moved to hospice care | 1
Not completed — technician error | 1
Not completed — Death | 3

BASELINE CHARACTERISTICS:
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.1 (10.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 28
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5
  Not Hispanic or Latino | 47
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 7
  White | 44
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 52

OUTCOME MEASURES:

1. Primary Outcome: Correlation of ⁸⁹Zr-Df-IAB22M2C Uptake in Biopsied Tumors With CD8+ Cell Measurement by Immunohistochemistry (IHC)
Description: Analyze ⁸⁹Zr-Df-IAB22M2C uptake in biopsied tumors as determined by SUV-based quantitative measures (SUVmax, SUVpeak, SUVmean, CD8 tumor volume, and tumor:reference tissue ratio) with CD8+ cell measurement determined by IHC from biopsy samples.
Time Frame: Baseline to 4-5 weeks after the start of immunotherapy
Population: Total number of patients with at least one evaluable biopsy sample and corresponding Zr-89 Df-AIB22M2C PET/CT scan
Measure: Number (95% Confidence Interval); unit: r
Groups:
- Renal Cell Carcinoma Subgroup: Subgroup of all participants enrolled with a diagnosis of Renal Cell Carcinoma who have at least one evaluable biopsy and corresponding 89Zr Df-IAB22M2C PET/CT scan
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion | Renal Cell Carcinoma Subgroup
Number analyzed (Participants) | 49 | 17
r | 0.3902 [0.1479 to 0.5751] | 0.7848 [0.5988 to 0.8650]

2. Primary Outcome: Number of Participants With Adverse Events
Description: Number of participants who experienced any treatment emergent adverse events
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
Participants | 40

3. Primary Outcome: Participants With Signs and Symptoms of Infusion Reactions
Description: Number of participants with reported signs or symptoms of infusion reactions
Time Frame: Up to 12 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
Participants | 0

4. Primary Outcome: Change in WBC Absolute Counts
Description: WBC absolute counts
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: For Treatment Visit 3, not all sites handle radioactive labs. For Treatment Visit 5, Fewer than 52 due to attrition. For Treatment Visit 6, not all sites handle radioactive labs. For Treatment Visit 7, only available for pts who attended for biopsy on-treatment For Treatment Visit 8, Fewer than 52 due to attrition.
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
10^9 cells/L
  Baseline | 7.6 (3.37)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 7.7 (3.96)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 6.3 (2.89)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 6.2 (1.67)
  Treatment Visit 7: number analyzed (Participants) | 20
  Treatment Visit 7 | 6.4 (3.07)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 6.4 (2.39)

5. Primary Outcome: Changes in Hematocrit (%) Laboratory Values
Description: hematocrit (%) laboratory values
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: % by volume of red cells
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
% by volume of red cells
  Baseline | 38.2 (5.44)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 37.7 (6.28)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 37.2 (4.86)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 38.7 (5.54)
  Treatment Visit 7: number analyzed (Participants) | 20
  Treatment Visit 7 | 36.6 (6.0)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 36.5 (5.87)

6. Primary Outcome: Changes in Hemoglobin (g/dL) Laboratory Values Compared With Baseline
Description: hemoglobin (g/dL) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: For Treatment Visit 3, not all sites handle radioactive labs. For Treatment Visit 5, Fewer than 52 due to attrition.
Measure: Mean (Standard Deviation); unit: g/dl
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
g/dl
  Baseline | 12.5 (2.52)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 12.4 (2.38)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 12.1 (2.44)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 12.8 (2.07)
  Treatment Visit 7: number analyzed (Participants) | 20
  Treatment Visit 7 | 12.1 (2.14)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 12.1 (2.06)

7. Primary Outcome: Changes in Platelet Count Laboratory Values Compared With Baseline
Description: platelet count laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
10^9 cells/L
  Baseline | 270.1 (136.33)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 224.5 (104.90)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 227.2 (105.01)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 227.0 (70.59)
  Treatment Visit 7: number analyzed (Participants) | 20
  Treatment Visit 7 | 249.7 (103.38)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 242.1 (93.42)

8. Primary Outcome: Changes in WBC Count Laboratory Values Compared With Baseline
Description: WBC count laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^9 cells/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
10^9 cells/L
  Baseline | 7.6 (3.37)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 7.7 (3.96)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 6.3 (2.89)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 6.2 (1.67)
  Treatment Visit 7: number analyzed (Participants) | 20
  Treatment Visit 7 | 6.4 (3.07)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 6.4 (2.39)

9. Primary Outcome: Changes in RBC Count Laboratory Values Compared With Baseline
Description: RBC count laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: 10^12 cells/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
10^12 cells/L
  Baseline | 4.3 (0.64)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 4.1 (0.81)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 4.2 (0.56)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 4.3 (0.68)
  Treatment Visit 7: number analyzed (Participants) | 20
  Treatment Visit 7 | 4.1 (0.63)
  Treatment Visit 8: number analyzed (Participants) | 4
  Treatment Visit 8 | 4.1 (0.70)

10. Primary Outcome: Changes in Blood Glucose (mg/dL) Laboratory Values Compared With Baseline
Description: blood glucose (mg/dL) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mg/dL
  Baseline: number analyzed (Participants) | 51
  Baseline | 115.986 (39.297)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 119.114 (39.447)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 115.534 (31.670)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 295.466 (580.168)
  Treatment Visit 7: number analyzed (Participants) | 18
  Treatment Visit 7 | 108.651 (17.977)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 113.208 (26.300)

11. Primary Outcome: Changes in Chloride Laboratory Values Compared With Baseline
Description: chloride laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: For Treatment Visit 3, not all sites handle radioactive labs. For Treatment Visit 5, Fewer than 52 due to attrition.
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mEq/L
  Baseline | 102.255 (3.903)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 102.769 (3.811)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 102.364 (3.498)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 103.900 (1.524)
  Treatment Visit 7: number analyzed (Participants) | 18
  Treatment Visit 7 | 103.059 (3.280)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 102.419 (2.905)

12. Primary Outcome: Changes in Potassium Laboratory Values Compared With Baseline
Description: Potassium laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mEQ/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mEQ/L
  Baseline: number analyzed (Participants) | 51
  Baseline | 4.314 (0.501)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 4.038 (0.386)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 4.223 (0.508)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 4.080 (0.452)
  Treatment Visit 7: number analyzed (Participants) | 18
  Treatment Visit 7 | 4.333 (0.351)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 4.233 (0.470)

13. Primary Outcome: Changes in Sodium Laboratory Values Compared With Baseline
Description: sodium laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mEq/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mEq/L
  Baseline: number analyzed (Participants) | 51
  Baseline | 137.510 (3.190)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 137.154 (1.908)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 137.227 (2.868)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 138.000 (1.764)
  Treatment Visit 7: number analyzed (Participants) | 18
  Treatment Visit 7 | 137.556 (2.854)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 137.326 (2.286)

14. Primary Outcome: Changes in Serum Creatinine (mg/dL) Laboratory Values Compared With Baseline
Description: serum creatinine (mg/dL) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mg/dL
  Baseline: number analyzed (Participants) | 51
  Baseline | 0.930 (0.289)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 0.958 (0.297)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 0.934 (0.332)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 0.961 (0.300)
  Treatment Visit 7: number analyzed (Participants) | 18
  Treatment Visit 7 | 0.834 (0.280)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 0.935 (0.353)

15. Primary Outcome: Changes in GGT (U/L) Laboratory Values Compared With Baseline
Description: GGT (U/L) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
U/L
  Baseline: number analyzed (Participants) | 23
  Baseline | 36.957 (36.921)
  Treatment Visit 3: number analyzed (Participants) | 10
  Treatment Visit 3 | 60.500 (80.845)
  Treatment Visit 5: number analyzed (Participants) | 21
  Treatment Visit 5 | 56.333 (79.741)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 77.700 (118.963)
  Treatment Visit 7: number analyzed (Participants) | 3
  Treatment Visit 7 | 17.333 (9.504)
  Treatment Visit 8: number analyzed (Participants) | 20
  Treatment Visit 8 | 88.200 (188.341)

16. Primary Outcome: Changes in BUN (mg/dL) Laboratory Values Compared With Baseline
Description: BUN (mg/dL) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mg/dL
  Baseline: number analyzed (Participants) | 50
  Baseline | 16.720 (7.600)
  Treatment Visit 3: number analyzed (Participants) | 12
  Treatment Visit 3 | 15.417 (5.452)
  Treatment Visit 5: number analyzed (Participants) | 43
  Treatment Visit 5 | 17.140 (6.947)
  Treatment Visit 6: number analyzed (Participants) | 9
  Treatment Visit 6 | 17.778 (7.259)
  Treatment Visit 7: number analyzed (Participants) | 17
  Treatment Visit 7 | 13.353 (5.219)
  Treatment Visit 8: number analyzed (Participants) | 42
  Treatment Visit 8 | 17.119 (9.868)

17. Primary Outcome: Changes in LDH (U/L) Laboratory Values Comapared With Baseline
Description: LDH (U/L) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
U/L
  Baseline: number analyzed (Participants) | 28
  Baseline | 236.821 (159.466)
  Treatment Visit 3: number analyzed (Participants) | 11
  Treatment Visit 3 | 281.000 (149.534)
  Treatment Visit 5: number analyzed (Participants) | 24
  Treatment Visit 5 | 310.375 (383.334)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 432.500 (417.848)
  Treatment Visit 7: number analyzed (Participants) | 3
  Treatment Visit 7 | 271.000 (133.907)
  Treatment Visit 8: number analyzed (Participants) | 24
  Treatment Visit 8 | 327.750 (369.221)

18. Primary Outcome: Total Bilirubin (mg/dL) Laboratory Values
Description: Total bilirubin (mg/dL) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mg/dL
  Baseline | 0.497 (0.279)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 0.562 (0.195)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 0.553 (0.325)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 0.511 (0.272)
  Treatment Visit 7: number analyzed (Participants) | 14
  Treatment Visit 7 | 0.559 (0.341)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 0.545 (0.306)

19. Primary Outcome: ALP Laboratory Values
Description: Change/shifts in ALP (U/L) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
U/L
  Baseline: number analyzed (Participants) | 50
  Baseline | 98.980 (46.687)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 111.000 (57.716)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 102.341 (61.689)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 123.400 (111.932)
  Treatment Visit 7: number analyzed (Participants) | 14
  Treatment Visit 7 | 97.357 (29.570)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 114.163 (112.280)

20. Primary Outcome: ALT Laboratory Values
Description: Change/shifts in ALT (U/L) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
U/L
  Baseline: number analyzed (Participants) | 50
  Baseline | 23.336 (17.428)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 25.615 (14.414)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 29.615 (22.315)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 37.700 (31.077)
  Treatment Visit 7: number analyzed (Participants) | 14
  Treatment Visit 7 | 27.071 (23.685)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 31.628 (34.590)

21. Primary Outcome: AST Laboratory Values
Description: Change/shifts in AST (U/L) laboratory values compared with baseline results.
Time Frame: Baseline, Visit 3 (Day 2), Visit 5 (Day 30-51) , Visit 6 (Day 31-52), Visit 7 (Day 30-65) and visit 8 (Day 58-86)
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
U/L
  Baseline: number analyzed (Participants) | 50
  Baseline | 25.740 (14.540)
  Treatment Visit 3: number analyzed (Participants) | 13
  Treatment Visit 3 | 32.769 (22.654)
  Treatment Visit 5: number analyzed (Participants) | 44
  Treatment Visit 5 | 31.932 (24.413)
  Treatment Visit 6: number analyzed (Participants) | 10
  Treatment Visit 6 | 50.700 (46.114)
  Treatment Visit 7: number analyzed (Participants) | 14
  Treatment Visit 7 | 23.143 (12.703)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 36.116 (35.116)

22. Primary Outcome: PR Interval Assessed by 12-Lead Electrocardiogram
Description: PR interval reported in milliseconds (msecs)
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51)
Population: fewer patients at later visits due to attrition
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
msec
  Baseline | 157.4 (30.97)
  Treatment visit 2 - 1 Hour Post Dose: number analyzed (Participants) | 50
  Treatment visit 2 - 1 Hour Post Dose | 159.1 (31.23)
  Treatment Visit 5 - Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5 - Pre Dose | 154.3 (25.55)
  Treatment Visit 5-1 Hour Post Dose: number analyzed (Participants) | 45
  Treatment Visit 5-1 Hour Post Dose | 159.2 (28.86)

23. Primary Outcome: Diastolic Blood Pressure
Description: Diastolic Blood Pressure
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51), Visit 8 (Day 58-86)
Population: Not all patients completed all timepoints.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
mmHg
  Baseline | 74.9 (8.94)
  Treatment Visit 2-Post Dose 1 Hour: number analyzed (Participants) | 49
  Treatment Visit 2-Post Dose 1 Hour | 74.1 (8.92)
  Treatment Visit 5-Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5-Pre Dose | 75.3 (7.26)
  Treatment Visit 5-Post Dose 1 Hour: number analyzed (Participants) | 44
  Treatment Visit 5-Post Dose 1 Hour | 74.9 (8.83)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 73.2 (8.65)

24. Primary Outcome: Evaluation of Heart Rate (Beats Per Minute)
Description: Changes/shifts in heart rate
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51), Visit 8 (Day 58-86)
Population: Not all patients completed all timepoints.
Measure: Mean (Standard Deviation); unit: beats/min
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
beats/min
  Baseline | 794 (12.30)
  Treatment Visit 2-Post Dose 1 Hour: number analyzed (Participants) | 49
  Treatment Visit 2-Post Dose 1 Hour | 75.6 (11.99)
  Treatment Visit 5-Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5-Pre Dose | 78.7 (13.90)
  Treatment Visit 5-Post Dose 1 Hour: number analyzed (Participants) | 44
  Treatment Visit 5-Post Dose 1 Hour | 76.5 (14.18)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 84.0 (17.49)

25. Primary Outcome: Evaluation of Respiration Rate
Description: Changes/shifts in respiration rate
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51), Visit 8 (Day 58-86)
Population: Not all patients completed all timepoints.
Measure: Mean (Standard Deviation); unit: breaths/min
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
breaths/min
  Baseline | 16.8 (2.78)
  Treatment Visit 2-Post Dose 1 Hour: number analyzed (Participants) | 49
  Treatment Visit 2-Post Dose 1 Hour | 17.2 (3.00)
  Treatment Visit 5-Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5-Pre Dose | 16.9 (2.28)
  Treatment Visit 5-Post dose 1 Hour: number analyzed (Participants) | 44
  Treatment Visit 5-Post dose 1 Hour | 16.7 (1.72)
  Treatment Visit 8: number analyzed (Participants) | 43
  Treatment Visit 8 | 17.1 (1.52)

26. Primary Outcome: Evaluation of Temperature
Description: Changes/shifts in temperature
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51), Visit 8 (Day 58-86)
Population: Not all patients completed all timepoints.
Measure: Mean (Standard Deviation); unit: degrees Celsius
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
degrees Celsius
  Baseline | 36.7 (0.30)
  Treatment Visit 2-Post Dose 1 Hour: number analyzed (Participants) | 49
  Treatment Visit 2-Post Dose 1 Hour | 36.7 (0.26)
  Treatment Visit 5-Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5-Pre Dose | 36.7 (0.30)
  Treatment Visit 5-Post Dose 1 Hour: number analyzed (Participants) | 44
  Treatment Visit 5-Post Dose 1 Hour | 36.7 (0.29)
  Treatment Visit 8: number analyzed (Participants) | 41
  Treatment Visit 8 | 36.6 (0.41)

27. Primary Outcome: QRS Interval Assessed by 12-Lead Electrocardiogram
Description: QRS Interval reported in milliseconds (msec)
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51)
Population: fewer patients at later visits due to attrition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
milliseconds
  Baseline: number analyzed (Participants) | 50
  Baseline | 89.7 (15.84)
  Treatment Visit 2: number analyzed (Participants) | 50
  Treatment Visit 2 | 90.4 (18.17)
  Treatment Visit 5 Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5 Pre Dose | 89.9 (16.47)
  Treatment Visit 5 Post Dose: number analyzed (Participants) | 45
  Treatment Visit 5 Post Dose | 90.5 (17.26)

28. Primary Outcome: QT Interval Assessed by 12-Lead Electrocardiogram
Description: QT interval reported in milliseconds (msec)
Time Frame: Baseline, Visit 2 (Day1), Visit 5 (Day 30-51)
Population: fewer patients at later visits due to attrition
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- ⁸⁹Zr-Df-IAB22M2C Infusion: A dose of 3 mCi (±20%) or 1mCi (±20%) ⁸⁹Zr-Df-IAB22M2C at 1.5 mg of API will be administered intravenously over 5-10 minutes, within one week prior to the onset of immunotherapy, and 5 to 6 weeks after start of IOT.
  ⁸⁹Zr-Df-IAB22M2C: ⁸⁹Zr-Df-IAB22M2C CD8 T cell tracer for Positron Emission Tomography (PET)
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
milliseconds
  Baseline | 387.6 (37.20)
  Treatment Visit 2: number analyzed (Participants) | 50
  Treatment Visit 2 | 394.0 (38.49)
  Treatment Visit 5 Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5 Pre Dose | 386.3 (39.87)
  Treatment Visit 5 Post Dose: number analyzed (Participants) | 45
  Treatment Visit 5 Post Dose | 398.3 (41.02)

29. Primary Outcome: QTc Interval Assessed by 12-Lead Electrocardiogram
Description: QTc interval reported in milliseconds (msecs)
Time Frame: Baseline, Visit 2 (Day 1), Visit 5 (Day 30-51)
Population: fewer patients at later visits due to attrition
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
milliseconds
  Baseline | 428.8 (24.92)
  Treatment Visit 2: number analyzed (Participants) | 50
  Treatment Visit 2 | 431.5 (24.49)
  Treatment Visit 5 Pre Dose: number analyzed (Participants) | 44
  Treatment Visit 5 Pre Dose | 430.3 (21.10)
  Treatment Visit 5 Post Dose: number analyzed (Participants) | 44
  Treatment Visit 5 Post Dose | 430.3 (21.10)

30. Secondary Outcome: Assessment of Baseline and On-treatment ⁸⁹Zr-Df-IAB22M2C Uptake and Distribution in Lymphoid Organs, and Measurement of Change Between the Paired Observations
Description: Assessment of Baseline and On-treatment ⁸⁹Zr-Df-IAB22M2C uptake and distribution in tumors and lymphoid organs, and measurement of change between the paired observations as determined by:
  -SUVs in reference tissues
Time Frame: 5 weeks
Measure: Mean (Full Range); unit: SUVmean
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
SUVmean
  Spleen baseline | 63.5 [23.7 to 113.9]
  Spleen on treatment | 58.7 [19.0 to 102.8]
  bone marrow baseline | 7.6 [4.2 to 13.0]
  bone marrow on treatment | 7.4 [2.8 to 15.9]

31. Secondary Outcome: Measurement of Change in ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) Uptake in Biopsied Tumors as Determined by SUV-based Quantitative Analysis
Description: Measurement of change in ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) uptake in biopsied tumors as determined by SUV-based quantitative analysis (e.g. SUVmax, SUVpeak, SUVmean)
Time Frame: 7 weeks
Population: 36 patients with evaluable PET-biopsy pairs at baseline 33 patients with evaluable PET-biopsy pairs at on treatment
Measure: Mean (Standard Deviation); unit: SUV
Groups:
- ⁸⁹Zr-Df-IAB22M2C Infusion: A dose of 3 mCi (±20%) or 1mCi (±20%) of ⁸⁹Zr-Df-IAB22M2C at 1.5 mg of API will be administered intravenously over 5-10 minutes, within one week prior to the onset of immunotherapy, and 5 to 6 weeks after start of IOT.
  ⁸⁹Zr-Df-IAB22M2C: ⁸⁹Zr-Df-IAB22M2C CD8 T cell tracer for Positron Emission Tomography (PET)
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
Number analyzed (Participants) | 52
SUV
  SUVmean baseline: number analyzed (Participants) | 36
  SUVmean baseline | 3.1 (3.2)
  SUVmax baseline: number analyzed (Participants) | 36
  SUVmax baseline | 5.1 (5.3)
  SUVpeak baseline: number analyzed (Participants) | 36
  SUVpeak baseline | 3.6 (4.2)
  SUVmean on treatment: number analyzed (Participants) | 33
  SUVmean on treatment | 4.0 (3.3)
  SUVmax on treatment: number analyzed (Participants) | 33
  SUVmax on treatment | 6.5 (5.0)
  SUVpeak on treatment: number analyzed (Participants) | 33
  SUVpeak on treatment | 4.6 (3.9)

32. Secondary Outcome: Description of Biodistribution Patterns of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) on PETbaseline and PETTx and Any Changes in Biodistribution Between Baseline and On-Treatment.
Description: Description of biodistribution patterns of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) on PETbaseline and PETTx and any changes in biodistribution between baseline and On-Treatment.
Time Frame: 7 weeks
Measure: Number; unit: number of lesions with this pattern
Units Other Than Participants: lesions
Groups:
- Lesions With Paired Values (i.e. Baseline and On-treatment Are Both Available) Are Included: Only lesions with paired values (i.e. CD8 PET/CT Baseline and On-treatment are both available) are included
Arm/Group | Lesions With Paired Values (i.e. Baseline and On-treatment Are Both Available) Are Included
Number analyzed (Participants) | 52
Number analyzed (lesions) | 69
number of lesions with this pattern
  Heterogeneous or Mixed -Heterogeneous or Mixed | 34
  Homogeneous - Heterogeneous or Mixed | 3
  Heterogeneous or Mixed - Homogeneous | 6
  Homogeneous - Homogeneous | 16
  Peripheral - Heterogeneous or Mixed | 2
  Peripheral - Peripheral | 8

33. Other Pre Specified Outcome: Correlation of Visual and Quantitative ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) Uptake in Tumor Lesions With Change in CD8+ T Cells as Determined by IHC From Biopsy Samples Obtained Prior to and 4 to 7 Weeks After the Start of Immunotherapy.
Description: Correlation of visual and quantitative ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) uptake in tumor lesions with change in CD8+ T cells as determined by IHC from biopsy samples obtained prior to and 4 to 7 weeks after the start of immunotherapy.
Time Frame: 7 weeks
Reporting Status: Not Posted

34. Other Pre Specified Outcome: Estimation of Positive Predictive Value, Negative Predictive Value, Sensitivity and Specificity of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) PET for Detecting CD8+ T Cells as Determined by IHC.
Description: Estimation of positive predictive value, negative predictive value, sensitivity and specificity of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) PET for detecting CD8+ T cells as determined by IHC.
Time Frame: 7 weeks
Reporting Status: Not Posted

35. Other Pre Specified Outcome: Assessment of Changes in ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) Uptake and Distribution From Baseline to 5-7 Days Start of Immunotherapy if Available.
Description: Assessment of changes in ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) uptake and distribution from baseline to 5-7 days start of immunotherapy if available.
Time Frame: 7 weeks
Reporting Status: Not Posted

36. Other Pre Specified Outcome: Correlation of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) Uptake With Clinical Outcomes (Response Rates, Duration of Response, Disease Stability Rate and PFS at Defined Intervals as Determined by the Local Investigator.
Description: Correlation of ⁸⁹Zr-Df-IAB22M2C (CD8 PET Tracer) uptake with clinical outcomes
Time Frame: 18 months
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 3 months
Description: AEs defined as any unfavorable or unintended sign, symptom, or disease that occurred or was reported by the patient, or a worsening of a pre-existing condition. Clinically significant lab results are regarded as AEs.
  Please note that most TEAEs are attributable to standard of care treatments rather than the study IP.
Arm/Group | ⁸⁹Zr-Df-IAB22M2C Infusion
All-Cause Mortality (participants affected / at risk) | 3/52
Serious Adverse Events (participants affected / at risk) | 11/52
Other Adverse Events (participants affected / at risk) | 40/52
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ⁸⁹Zr-Df-IAB22M2C Infusion (N=52)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Diarrhoea (Gastrointestinal disorders) | 1 (1)
Large intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1)
Pneumonia (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Compression fracture (Injury, poisoning and procedural complications) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Intracardiac thrombus (Cardiac disorders) | 1 (1)
Asthenia (General disorders) | 1 (1)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Acidosis (Metabolism and nutrition disorders) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ⁸⁹Zr-Df-IAB22M2C Infusion (N=52)
Constipation (Gastrointestinal disorders) | 8 (8)
Nausia (Gastrointestinal disorders) | 7 (11)
Diarrhoea (Gastrointestinal disorders) | 6 (13)
Vomiting (Gastrointestinal disorders) | 6 (8)
Abdominal pain (Gastrointestinal disorders) | 5 (5)
Dry mouth (Gastrointestinal disorders) | 3 (4)
Abdominal distension (Gastrointestinal disorders) | 2 (2)
Fatigue (General disorders) | 8 (9)
Pyrexia (General disorders) | 4 (5)
Oedema peripheral (General disorders) | 3 (5)
Chills (General disorders) | 2 (2)
Pain (General disorders) | 2 (2)
Hypokalaemia (Metabolism and nutrition disorders) | 6 (9)
Decreased appetite (Metabolism and nutrition disorders) | 6 (7)
Dehydration (Metabolism and nutrition disorders) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 3 (3)
Hypomansesaemia (Metabolism and nutrition disorders) | 2 (3)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hyponatraemia (Metabolism and nutrition disorders) | 2 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (6)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Pruritis (Skin and subcutaneous tissue disorders) | 8 (9)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 (2)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 (7)
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (3)
Blood creatinine increased (Investigations) | 3 (5)
Aspartate aminotransferase increased (Investigations) | 2 (4)
Alanine aminotransferase increased (Investigations) | 2 (3)
Gamma-glutamyltransferase increased (Investigations) | 2 (3)
Weight decreased (Investigations) | 2 (3)
Lymphocyte count decreased (Investigations) | 2 (2)
Hypertension (Vascular disorders) | 6 (34)
Hypotension (Vascular disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 4 (6)
Procedural pain (Injury, poisoning and procedural complications) | 3 (3)
Contusion (Injury, poisoning and procedural complications) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 4 (5)
Anxiety (Psychiatric disorders) | 3 (5)
Insomnia (Psychiatric disorders) | 3 (3)
Headache (Nervous system disorders) | 2 (2)
Anaemia (Blood and lymphatic system disorders) | 3 (7)
Thrompocytopenia (Blood and lymphatic system disorders) | 3 (3)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (3)
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-28): https://cdn.clinicaltrials.gov/large-docs/23/NCT03802123/Prot_SAP_000.pdf